CLINICAL TRIAL: NCT03755635
Title: Neonatal Sepsis at Neonatal Intensive Care Units of Two Major Referral Hospitals in Ghana
Brief Title: Neonatal Sepsis at Neonatal Intensive Care Units in Ghana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stephanie Bjerrum (Other)
Collaborators: University of Copenhagen (Other); Korle-Bu Teaching Hospital, Accra, Ghana (Other); Rigshospitalet, Denmark (Other); University of Ghana (Other)
Responsible Party: Sponsor-Investigator, Stephanie Bjerrum, MD, PHD, postdoc, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UM ID: 892333
Record Dates: First submitted 2018-11-23; First posted 2018-11-28 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Neonatal SEPSIS
Keywords: Neonatal sepsis; Infection control; Hand hygiene; WHO multi modal
MeSH Terms: conditions — Neonatal Sepsis | interventions — Hand Hygiene

STUDY DESIGN:
Intervention Model Description: Controlled before and after interventional trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Continuously monitoring of neonatal sepsis under standard of care at one site
- Hand hygiene (Experimental): The WHO multimodal hand hygiene strategy is implemented at one site
  Interventions: Combination Product: The WHO multimodal hand hygiene strategy

INTERVENTIONS:
Combination Product: The WHO multimodal hand hygiene strategy — Comprises five essential elements; system change-availability of alcohol-based hand rub at the point of care and/ or access to safe continuous water supply and soap and towels; training and education of healthcare professionals; monitoring of hand hygiene practices and performance feedback; reminders in the workplace; and the creation of a hand hygiene safety culture with the participation of both individual healthcare workers and senior hospital managers.
  Other Names: Hand hygiene
  Arms: Hand hygiene

SUMMARY:
Background: Neonatal sepsis is a major contributor to global under five mortality. In developing countries a major proportion of neonatal sepsis is thought to emanate from the healthcare setting, due to challenges in infection prevention practices.

Aim: To study the epidemiology of neonatal sepsis and evaluate the effect of multimodal infection control interventions on the incidence of neonatal sepsis; and colonization by multidrug resistant Gram negative bacteria (MDRGNB).

Methods: A controlled before and after interventional trial comprising a 7 month pre- intervention phase, 5 month intervention phase and 7 month post-intervention phase. Neonates admitted at the Neonatal Intensive Care Unit (NICU) at Korle-Bu Teaching Hospital (KBTH) will be enrolled prospectively and followed up for diagnosis of sepsis and outcome of admission. This will be used to describe the epidemiology of neonatal sepsis. Swabs will be collected from a subpopulation of included neonates at intervention site (KBTH) and control site (37 Military Hospital) NICUs to assess colonization of neonates with MDRGNB. Environmental swabs will be collected from surfaces at the NICU to assess MDRGNB contamination of the environment. The intervention comprises infection prevention strategies including implementation of the WHO multimodal hand hygiene strategy. The primary endpoint is incidence of neonatal sepsis.

Expected Outcome: This study will contribute to improved infection prevention practices in the participating NICUs and highlight lessons which other national and regional NICUs may learn from.

DETAILED DESCRIPTION:
Background In 2012, it was estimated that approximately 680,000 neonatal deaths in developing countries were due to bacterial infections, with an incidence risk of 7.6% and a case fatality risk of 9.8. A major proportion of neonatal infections are expected to be health-care associated, due to inadequate infrastructure and resources for infection control and prevention. Hospital acquired infections(HAIs) are associated with multi-drug resistant (MDR) bacteria, which increases the risk of therapeutic failure due to the limited choice of available antibiotics. HAIs also lead to extended duration of admission, increased medical costs, morbidity and mortality.

Transmission of MDR bacteria in the hospital environment is thought to be due to unhygienic practices which occur during clinical invasive procedures, (e.g. artificial ventilation, catheter and intravenous line insertion). Neonatal infections may also be due to invasion by colonizing bacteria of the neonate, usually originating from maternal and environmental flora.

According to the WHO, 50% of HAIs are preventable through implementation of infection control practices. The WHO has instituted a multimodal hand hygiene strategy that has been found to improve hand hygiene compliance and reduce the prevalence of HAIs. However, the effectiveness of this strategy in a neonatal intensive care unit (NICU) with high risk of colonization with environmental bacteria has not been studied. In fact, most studies that have examined the potential sources and mode of transmission of organisms that cause neonatal sepsis have been conducted in well-resourced countries.

The hypothesis of the study is that the hospital environment serves as a source of MDR Gram negative bacteria responsible for neonatal colonization and sepsis among patients admitted at the NICU of the KBTH; and that implementation of the multimodal hand hygiene strategy will lead to a reduction in the incidence of neonatal sepsis and colonization by MDR Gram negative bacteria.

Objective To determine the impact of multi-modal infection control interventions on the incidence of neonatal sepsis and colonization by MDR Gram negative bacteria.

Method This study will evaluate the impact of WHO multimodal hand hygiene strategy on the incidence of neonatal sepsis and neonatal colonization by MDR Gram negative bacteria as well as pilot surveillance of neonatal sepsis at the participating sites.

Study setting: Data will be collected at the NICU of the KBTH and the 37 Military Hospital, Accra, Ghana.

Study Design: The study will be a controlled before and after interventional trial with one interventional site (KBTH) and a control site (37 Military hospital). Data will be collected over 19 months with a baseline phase of 7 months; an interventional phase of 5 months; and a post intervention phase of 7 months.

Intervention: The WHO multimodal hand hygiene strategy comprises five essential elements; system change-availability of alcohol-based hand rub at the point of care and/ or access to safe continuous water supply and soap and towels; training and education of healthcare professionals; monitoring of hand hygiene practices and performance feedback; reminders in the workplace; and the creation of a handhygiene safety culture with the participation of both individual healthcare workers and senior hospital managers.

ELIGIBILITY:
Inclusion Criteria:

* Admission NICU
* Birth weight ≥750 Grams
* ≤48 hours of age at time of enrolment
* Consent to participate obtained from legal guardian

Exclusion Criteria:

* Neonates with severe congenital malformations
* Neonates who have undergone surgical procedure

Ages: 1 Minute to 48 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5433 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of neonatal sepsis | Post-intervention at 7 months
  Incidence of neonatal sepsis including clinical cases treated as sepsis and cases of neonatal sepsis with confirmed bloodstream infections per 1000 admissions.

SECONDARY OUTCOMES:
Rate of hand hygiene compliance per opportunity | Post-intervention at 7 months
  Hand hygiene events per opportunity for hand hygiene measured by direct observations
Rate of MDR Gram negative bacteria colonization among neonates | During intervention at 2 months and post-intervention at 7 months
  Prevalence of MDR Gram negative bacteria among admitted neonates
Length of admission in days | Post-intervention at 7 months
  Days of admission
All-cause mortality | Post-intervention at 7 months
  Mortality rates during admission

CONTACTS AND LOCATIONS:
Overall Officials: Appiah Korang Labi, MD, Principal Investigator — Department of Int. Health and Immunlogy Microbiology, University og Copenhagen; Jørgen Kurtzhals, Professor, Study Director — Department of Int. Health and Immunlogy Microbiology, University og Copenhagen
Locations (1):
- Korle Bu Teaching Hospital, Accra, Ghana

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Labi AK, Enweronu-Laryea CC, Nartey ET, Bjerrum S, Ayibor PK, Andersen LP, Newman MJ, Kurtzhals JAL. Bloodstream Infections at Two Neonatal Intensive Care Units in Ghana: Multidrug Resistant Enterobacterales Undermine the Usefulness of Standard Antibiotic Regimes. Pediatr Infect Dis J. 2021 Dec 1;40(12):1115-1121. doi: 10.1097/INF.0000000000003284. PMID 34561387